CLINICAL TRIAL: NCT03959826
Title: Promoting Employment in Persons Living With HIV/AIDS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Carla Rash, Assistant Professor, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-178-2
Record Dates: First submitted 2019-05-17; First posted 2019-05-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Unemployment; HIV
Keywords: contingency management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Job activity contracting (Active Comparator): Standard services plus job activity contracting
  Interventions: Behavioral: activity contracting
- Reinforcement for completing activities (Experimental): Standard services plus job activity contracting plus reinforcement for completing job-related activities
  Interventions: Behavioral: activity contracting; Behavioral: contingency management for activity completion

INTERVENTIONS:
Behavioral: activity contracting — Participants will complete job-related activity contracts each week with the goal of obtaining employment.
Behavioral: contingency management for activity completion — Participants will earn chances to win prizes for completing specific job-related activities.
  Arms: Reinforcement for completing activities

SUMMARY:
Many persons living with HIV/AIDS (PLWHA) are unemployed, with estimates indicating rates as high as 60%. This study will examine the efficacy of reinforcing job-acquisition activities for improving employment outcomes in PLWHA who desire to return to the workforce in part- or full-time capacity. In total, this study will randomly assign 144 unemployed PLWHA to one of two interventions. All participants will receive usual unemployment services with an emphasis on specific issues related to HIV/AIDS, plus encouragement for completing activities geared toward employment readiness and acquisition. The enhanced intervention will involve that same treatment plus chances to win prizes for engaging in job-related activities each week. Participants will receive study treatments for 16 weeks and complete follow-up evaluations throughout 18 months. The hypothesis is that participants reinforced for completing job-related activities will transition to employment at higher and faster rates and work more often than those who are not reinforced for job-related activities.

DETAILED DESCRIPTION:
Many persons living with HIV/AIDS (PLWHA) are unemployed, with estimates indicating rates as high as 60%. This study will examine the efficacy of reinforcing job-acquisition activities for improving employment outcomes in PLWHA who desire to return to the workforce in part- or full-time capacity. In total, this study will randomly assign 144 unemployed PLWHA to one of two interventions. All participants will receive usual unemployment services with an emphasis on specific issues related to HIV/AIDS, plus encouragement for completing activities geared toward employment readiness and acquisition. The enhanced intervention will involve that same treatment plus chances to win prizes for engaging in job-related activities each week. Participants will receive study treatments for 16 weeks and complete follow-up evaluations throughout 18 months. Structured evaluations will assess employment outcomes, quality of life indices, physical and cognitive functioning, psychological symptoms, viral loads, and drug use and risk behaviors. The hypothesis is that participants reinforced for completing job-related activities will transition to employment at higher and faster rates and work more often than those who are not reinforced for job-related activities. The investigators also expect the reinforcement intervention will increase quality of life, reduce depressive symptoms, and improve medical outcomes. Compared to the standard care condition, it may also maintain or improve cognitive functioning and medication adherence and reduce risk behaviors that spread infectious diseases. The investigators will evaluate moderators and mediators of key employment and health outcomes, with an emphasis on exploring the extent to which work conditions (temporary, under the table, physically or emotionally demanding jobs etc.) impact psychosocial and physical health.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* aged 18+ years
* not working in the formal economy

Exclusion Criteria:

* have a condition that may hinder study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-06-12 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
job attainment | 18 months
  self-report of job attainment: yes/no
proportion of days worked for pay | 18 months
  self-report of number of days worked

CONTACTS AND LOCATIONS:
Overall Officials: Carla Rash, Ph.D., Principal Investigator — UConn Health
Locations (1):
- United Labor Agency, Middletown, Connecticut, United States